CLINICAL TRIAL: NCT06362070
Title: Comparison of Outcomes of Multiple Platforms for Assisted Robotic - Gastrectomy (COMPAR-G) in Gastric Cancer Patient.
Brief Title: Comparison of Outcomes of Multiple Platforms for Assisted Robotic - Gastrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMPAR-G
Record Dates: First submitted 2024-04-03; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Gastric Cancer; Gastrointestinal Cancer; Neoplasms; Gastric Diffuse Adenocarcinoma; Gastric Neoplasm; Stomach Adenocarcinoma
Keywords: Robotic-assisted surgery; Multiple surgical platforms; Postoperative complications; Operative outcomes; Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms; Gastrointestinal Neoplasms; Neoplasms; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- DaVinci® Surgical System (Active Comparator): Robot-assisted total or subtotal Gastrectomy is carried out through daVinci platform.
  (10 patients enrolled for phase 1 of the study and 15 patients for phase 2)
  Interventions: Device: DaVinci® Surgical System
- Hugo™ RAS System (Experimental): Robot-assisted total or subtotal Gastrectomy is carried out through Hugo platform.
  (10 patients enrolled for phase 1 of the study and 15 patients for phase 2)
  Interventions: Device: Hugo™ RAS System
- Versius® Robotic Surgery System (Experimental): Robot-assisted total or subtotal Gastrectomy is carried out through Versius platform.
  (10 patients enrolled for phase 1 of the study and 15 patients for phase 2)
  Interventions: Device: Versius® Robotic Surgery System

INTERVENTIONS:
Device: DaVinci® Surgical System — Assisted-robotic radical Gastrectomy
  Arms: DaVinci® Surgical System
Device: Hugo™ RAS System — Assisted-robotic radical Gastrectomy
  Arms: Hugo™ RAS System
Device: Versius® Robotic Surgery System — Assisted-robotic radical Gastrectomy
  Arms: Versius® Robotic Surgery System

SUMMARY:
The object of this exploratory clinical trial is to evaluate intra and post-operative complications in a population that underwent Robotic Gastrectomy, with multiple platforms:

* DaVinci;
* Hugo;
* Versius.

This study is divided into two phases: in the first phase, gastrectomy will be performed using both the new platforms (Hugo and Versius) and the standard platform (Da Vinci), to evaluate the feasibility of the surgical procedure. In the second phase, the three platforms will be compared to evaluate any differences in the learning curve for an upper-GI surgeon, expert in laparoscopic surgery but not with robotic one.

The questions it aims to answer are:

* Are differences (intra-operative, post-operative, oncological, functional, technical, and economic) among the three different platforms observable?
* Are there any differences between the three platforms related to the learning curve for surgeons?

Participants will be enrolled, after obtaining informed consent, in one of the following cohorts:

1. surgery with the daVinci platform;
2. surgery with the Hugo platform;
3. surgery with the Versius platform.

DETAILED DESCRIPTION:
Gastrectomy for gastric cancer could be performed through open, laparoscopic and robotic approaches. In the last ten years, robotic surgery, performed with Da Vinci® Robotic System (Intuitive Surgical Inc., Sunnyvale, CA, USA) has been introduced and increasingly used globally also in the field of gastric surgery. Indeed, the technological implementation obtained with the use of robotic surgery should guarantee an easier approach to the different phases of gastric surgery, and in particular to the more complex steps relating to the reconstructive phase of the operation.

Recently, after Intuitive patent expiration, two new CE-marked robotic platforms are available in Europe for minimally invasive procedures:

* Versius® Robotic Surgery System, (Cambridge Medical Robotics (CMR) Ltd., Cambridge, UK);
* HugoTM RAS (Medtronic Dublin, Ireland; Minneapolis, MN, USA).

Both platforms are currently used for urological and gynecological procedures, but, no experiences are reported in Literature related to the field of oncological esophago-gastric surgery. In order to provide evidence regarding the new robotic platforms, the COMPAR-G study has been designed to directly compare the Da Vinci® (as standard), Versius® and HugoTM RAS robotic platforms during gastrectomy.

In this regard, this study was proposed, divided into two phases: a first phase for feasibility of surgical procedure with different platforms and the second one to evaluate the learning curve for surgeons.

This second phase will be carried out only in the event of an extension of the rental of the two new platforms for a further period of one year.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 80 years
* Informed consent provided
* Primary stomach tumor
* Total or subtotal gastrectomy
* Tumour stage: T1-4a, any N, M0
* ASA I-III
* No BMI limits
* Upfront surgery or after neoadjuvant chemotherapy

Exclusion Criteria:

* Extension to esophagectomy
* Tumor of the esophago-gastric junction (Siwert I-III)
* Emergency surgery
* Metastatic patients (stage IV)
* Patients undergoing preoperative radiotherapy
* Previous major supramesocolic surgery (excluding cholecystectomy)
* Other coexisting malignant neoplasms

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Conversion rate to open or laparoscopic approach (Phase 1) | Intraoperative
  Number of procedures in which it is necessary to convert to open or laparoscopic approach, due to surgical and/or oncological needs
Number of participants with major intraoperative complications (Phase 1) | Intraoperative
  Major complications are considered according to the GASTRODATA definition (Unintentional intraoperative damage to major vessels and/or organs requiring reconstruction or resection. Intraoperative bleeding requiring urgent treatment. Unforeseen medical conditions that interrupt or change the planned procedure) and according to Clavien-Dindo Classification (7 grades: I, II, IIIa, IIIb, IVa, IVb and V): the higher the grade, the higher the severity of the complication.
Evaluation of surgical times of the standardized procedures (Phase 2) | Intraoperative
  Analysis of surgical times (as minutes of the different surgical steps of the standardized procedure).
Analysis of video of surgical procedures (Phase 2) | Intraoperative
  Evaluation of analysis of video of surgical procedure, as deviations from the standard.

SECONDARY OUTCOMES:
Estimated Blood Loss | Intraoperative
  Volume of blood loss (ml)
Overall duration of the surgery | Intraoperative
  Minutes
Anesthesia, Lymphadenectomy, Gastrectomy (10 different surgical steps) | Entrance of patient into operating room until completion of surgery
  Minutes
Number of participants with major postoperative complications | Until 90 days post surgery
  Major complications are considered according to GASTRODATA definition (surgical and/or general) and according to Clavien-Dindo Classification (7 grades: I, II, IIIa, IIIb, IVa, IVb and V): the higher the grade, the higher the severity of the complication
Compliance rate to ERAS protocol | 1-7 days postoperative
  Adherence to Enhanced recovery after surgery for gastric cancer (ERAS-GC) protocol, which involves a rapid mobilisation and refeeding of patiens.
Postoperative hospitalization | From the surgery day up to 20 days postoperative
  Days of recovery until the date of release
Postoperative pain | 1-5 days postoperative
  Numerical Rating Scale (NRS) 0-10 scale for the self-reported rate of pain: zero meaning "no pain" and 10 meaning "the worst pain imaginable"
Re-admission rate to hospitalization | Up to 90 days postoperative
  Number of patients readmitted to the hospital for postoperative complications
Damage due to positioning | Intraoperative
  Number of damage due to positioning on the operating bed, during the surgical procedure
Positive Surgical Margin | Up to 2 weeks postoperative (during histological analysis)
  Positive margin (distal or proximal) at histological examination
Lymph nodes resection | Up to 2 weeks postoperative (during histological analysis)
  Number of lymph nodes removed
Quality of Life Evaluation | Postoperaive (follow up at 1 month)
  EORTC QLQ-C30 questionnaire (30-item instrument designed to measure quality of life in all cancer patients) and EORTC STO-22 questionnaire (for measuring the QOL of patient with gastric cancer)
Time taken for platform-related technical steps | From the room setting, through surgical procedure until postoperative room restoration for each of expected surgeries
  Set up of operating table, Electric connections, Draping, Undraping, Docking, Undocking, Cleaning: time in minutes
Possible malfunction of the platform | Intraoperative
  Note
Non-Technical Skills Assessment (NTS) demonstrated by members of the surgical team during the intraoperative phase. | Intraoperative
  Targeted observation with "I.C.A.R.S" checklist (Interpersonal and Cognitive
  Assessment for Robotic Surgery) which includes following domains:
  Checklist and equipment; Interpersonal skills and Cognitive skills.
Procedure-related costs | From surgical procedure up to 90 days after surgery
  Estimate

CONTACTS AND LOCATIONS:
Locations (1):
- General and Upper GI Unit, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haig F, Medeiros ACB, Chitty K, Slack M. Usability assessment of Versius, a new robot-assisted surgical device for use in minimal access surgery. BMJ Surg Interv Health Technol. 2020 May 22;2(1):e000028. doi: 10.1136/bmjsit-2019-000028. eCollection 2020. PMID 35047788
- [Result] Peters BS, Armijo PR, Krause C, Choudhury SA, Oleynikov D. Review of emerging surgical robotic technology. Surg Endosc. 2018 Apr;32(4):1636-1655. doi: 10.1007/s00464-018-6079-2. Epub 2018 Feb 13. PMID 29442240
- [Result] Solaini L, D'Ignazio A, Marrelli D, Marano L, Avanzolini A, Morgagni P, Roviello F, Ercolani G. The effect of learning curve on perioperative outcomes of robotic gastrectomy in two western high-volume centers. Int J Med Robot. 2021 Apr;17(2):e2212. doi: 10.1002/rcs.2212. Epub 2021 Jan 8. PMID 33340239
- [Result] Li Z, Qian F, Zhao Y, Chen J, Zhang F, Li Z, Wang X, Li P, Liu J, Wen Y, Feng Q, Shi Y, Yu P. A comparative study on perioperative outcomes between robotic versus laparoscopic D2 total gastrectomy. Int J Surg. 2022 Jun;102:106636. doi: 10.1016/j.ijsu.2022.106636. Epub 2022 Apr 26. PMID 35472517
- [Result] Shibasaki S, Suda K, Hisamori S, Obama K, Terashima M, Uyama I. Robotic gastrectomy for gastric cancer: systematic review and future directions. Gastric Cancer. 2023 May;26(3):325-338. doi: 10.1007/s10120-023-01389-y. Epub 2023 Apr 3. PMID 37010634
- [Result] Prata F, Ragusa A, Tempesta C, Iannuzzi A, Tedesco F, Cacciatore L, Raso G, Civitella A, Tuzzolo P, Calle P, Pira M, Pino M, Ricci M, Fantozzi M, Prata SM, Anceschi U, Simone G, Scarpa RM, Papalia R. State of the Art in Robotic Surgery with Hugo RAS System: Feasibility, Safety and Clinical Applications. J Pers Med. 2023 Aug 6;13(8):1233. doi: 10.3390/jpm13081233. PMID 37623483
- [Result] Baiocchi GL, Giacopuzzi S, Marrelli D, Reim D, Piessen G, Matos da Costa P, Reynolds JV, Meyer HJ, Morgagni P, Gockel I, Lara Santos L, Jensen LS, Murphy T, Preston SR, Ter-Ovanesov M, Fumagalli Romario U, Degiuli M, Kielan W, Monig S, Kolodziejczyk P, Polkowski W, Hardwick R, Pera M, Johansson J, Schneider PM, de Steur WO, Gisbertz SS, Hartgrink H, van Sandick JW, Portolani N, Holscher AH, Botticini M, Roviello F, Mariette C, Allum W, De Manzoni G. International consensus on a complications list after gastrectomy for cancer. Gastric Cancer. 2019 Jan;22(1):172-189. doi: 10.1007/s10120-018-0839-5. Epub 2018 May 30. PMID 29846827